CLINICAL TRIAL: NCT02464852
Title: Assessment of the Effects of Sheffield Support Snood in MND Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STH18733
Record Dates: First submitted 2015-04-23; First posted 2015-06-08 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2015-06

CONDITIONS: Motor Neurone Disease
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Head Movements; Activities of Daily Living; Drinking; Hand Disinfection; Eating

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Snood (Other): All recruited participants will try out the snood
  Interventions: Behavioral: Head movements; Behavioral: Activities of daily living (drinking, washing hand and eating); Device: Sheffield Support Snood; Device: sEMG

INTERVENTIONS:
Behavioral: Head movements — Participants will be asked to perform a series of movements of exploration of their maximum neck range of motion, including: flexion, extension, right and left lateral flexion, right and left axial rotation.
Behavioral: Activities of daily living (drinking, washing hand and eating) — Patients will be asked to perform a series of activities of daily living (drinking, eating and washing hands).
Device: Sheffield Support Snood
Device: sEMG

SUMMARY:
The aim of this study is to evaluate the effects on MND patients of a new collar specifically designed for people affected by neck weakness: the Sheffield Support Snood.

DETAILED DESCRIPTION:
Motor Neurone Disease (MND) is neurodegenerative disorder that leads to progressive weakness of limb, bulbar and respiratory muscles. The most common form of the disease is the Amyotrophic Lateral Sclerosis (ALS). Severe weakness of the neck extensor muscles is common in patients with ALS. Those patients are advised to wear a cervical collar, to improve their neck posture and social interaction. However the main limit of commercially available collars is that they are designed to immobilize the neck, which makes them uncomfortable and strenuous to wear for long time. The aim of this study is to evaluate the effects on MND patients of a new collar specifically designed for people affected by neck weakness: the Sheffield Support Snood. The assessment will be performed through the use of inertial sensors since they allow the measurement to be performed in real life settings (clinics/home) with reduced discomfort to the patient. Subjects will be asked to perform a series of active head movements (flexion, extension, axial rotation, lateral bending) with and without the collar and the range of movement measured in the two cases will be used to assess the support offered by the collar. Since in MND patients difficulty in perform active head movements is due to a severe weakness of the extensor muscles, with or without involvement of the neck flexors, this study will also investigate the activation of these muscles while the subject is performing the active head movements. A wireless surface electromyographic system (sEMG) will be used to this purpose. Patients able to perform a series of activities of daily living (ADL, ie: drinking, eating, washing hands) will be asked to perform the tasks both with and without the collar. The support perceived by the subjects while they are performing the ADL will be evaluated through a questionnaire specifically developed for this study.

ELIGIBILITY:
Inclusion Criteria:

* Clinical status consistent with MND
* Capability to understand instructions
* Capability to perform testing procedures
* Ability to give informed consent

Exclusion Criteria:

* Presence of any inflammatory or other disease involving joint or muscle pathology that might affects testing results
* Unable to give informed consent

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-04; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
angular velocity and acceleration measured by the inertial sensors | while the subject is performing the head movements (Extension, flexion, axial rotation and lateral bending). Data collection will take approximately 30 minutes
electrical activity produced by the muscle measured by the EMG system | while the subject is performing the head movements (Extension, flexion, axial rotation and lateral bending). Data collection will take approximately 30 minutes
Description of the support perceived. It will be evaluated through a questionnaire which will include a series of sentences that describe the support offered by the collar. The subjects will be asked to state how much they agree with those sentences. | after the subject has performed the head movements (Extension, flexion, axial rotation and lateral bending). Answer the questionnaire will take approximately 10 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Hallamshire Hospital, Sheffield, South Yorkshire, United Kingdom